CLINICAL TRIAL: NCT00782262
Title: Effects of Obesity and Diet Induced Weight Loss on Cardiovascular Risk Factors, Vascular and Ventricular Structure and Function in Obese Men
Brief Title: Weight Loss Effects on Heart and Blood Vessel Function in Obesity
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Adelaide (Other)
Collaborators: Royal Adelaide Hospital (Other)
Responsible Party: Dr Cynthia Piantadosi, University of Adelaide and Royal Adelaide Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 050226
Record Dates: First submitted 2008-10-28; First posted 2008-10-31 (Estimated); Last update posted 2008-10-31 (Estimated); Status verified 2008-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (n=20) (Other): BP < 140/90, no diabetes mellitus and fasting glucose < 5.5
  Interventions: Dietary Supplement: KicStart™
- Group 2 (n=20) (Other): BP > 140/100, no diabetes mellitus and fasting glucose < 5.5
  Interventions: Dietary Supplement: KicStart™
- Group 3 (n=20) (Other): BP <140/100, no diabetes mellitus, fasting glucose 5.5 - 6.9
  Interventions: Dietary Supplement: KicStart™

INTERVENTIONS:
Dietary Supplement: KicStart™ — KicStart™ is a nutritionally complete, but lower energy formulated liquid meal. Two sachets of KicStart™ (one for breakfast and one for lunch) provides 450 cal of energy per day, 0.8 grams per kilogram ideal body weight of high quality protein, and the recommended daily allowances (RDI) of minerals, vitamins, trace elements, omega 3 and 6 essential fatty acids. The Kicstart is supplemented with some salads, carbohydrate free vegetables and a small piece of meat fish or chicken each day in order to achieve a total energy intake of approximately 850 kcals/day.

SUMMARY:
Obesity is a growing epidemic and is associated with an increased risk of heart attack and stroke. The investigators know that obesity leads to abnormalities in how the blood vessels and the heart function and that these abnormalities are an important cause of this increased risk in obese individuals. While improvements in these abnormalities have been reported with marked weight reduction (eg surgery) and lifestyle changes including exercise training, it is not clear that these abnormalities can be substantially reversed with standard dietary interventions. Additional information is needed regarding the degree of weight loss required, the time course of these improvements, nor the mechanisms. All of these have major implications for the potential role of weight loss in the management of these patients.

The investigators will assess the effects of dietary induced weight loss in both the short and long term on the function of blood vessels and the heart, and the relationship of any changes with markers of inflammation that are present in obesity.

By understanding the factors that are important in reversing these abnormalities in obesity the investigators will be better to identify and reduce heart attack and stroke in obese individuals in the future.

ELIGIBILITY:
Inclusion Criteria:

* Obese Caucasian men age 18-65 years, who are non smokers, and consuming 2 or fewer standard alcoholic drinks per day (on average over the past 5 years) will be recruited.
* Obesity, for the purposes of this study, is defined by a BMI > 30 and a waist circumference > 102 cm.
* Caucasian men only are enrolled because the cut-off points for the definition of obesity vary significantly by race.

Exclusion Criteria:

* Men are excluded if they have any previously diagnoses or symptomatic atherosclerotic disease, or are taking any cardiovascular medication.
* Men with known gallstones, history of gout, or any contraindication to MRI are also excluded.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2005-04; Primary Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
This will be the first analysis of the impact of rapid aggressive weight loss in obese individuals on both short and long-term cardiovascular indices. | 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Adelaide, Royal Adelaide Hospital, Adelaide, South Australia, Australia